CLINICAL TRIAL: NCT00488293
Title: Impact of Teledermatology on Health Services Outcomes in the VA
Brief Title: Impact of Teledermatology on Health Services Outcomes in the Department of Veterans Affairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 05-278
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Skin Diseases; Telemedicine; Quality of Life
Keywords: Telemedicine; Skin diseases; Dermatology; Quality of life; Economics
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Store and forward teledermatology consult process
  Interventions: Procedure: Store and forward teledermatology
- Arm 2 (No Intervention): Conventional consult process

INTERVENTIONS:
Procedure: Store and forward teledermatology — Standard electronic consult, standardized history, and image set
  Other Names: Teledermatology
  Arms: Arm 1

SUMMARY:
This study compares store and forward teledermatology with the conventional clinic-based consult process. Our primary objective is to determine whether the mean change in quality of life, as rated by the subscale scores and composite score on the Skindex-16 differs between the store and forward and conventional care modalities.

DETAILED DESCRIPTION:
Anticipated Impact on Veterans' Healthcare - Teledermatology has the potential to have a significant impact on veterans' healthcare. There is an unmet demand for Dermatology services distributed throughout a nation-wide patient base. Decentralization of care through the expansion of Community Based Outpatient Centers (CBOCs) adds to the demand for these services. Dermatologic care typically resides only at the largest medical centers within a Veterans Integrated Service Network (VISN). Teledermatology is one means of meeting the demand for Dermatology services by delivering dermatologic care to those sites that are geographically removed from the Dermatology Consult Service.

Project Background - For the majority of ambulatory skin conditions encountered in Primary Care and Dermatology Clinics the impact those conditions have on patients' quality of life is of principal importance. Commonly encountered skin diseases frequently result in discomfort or pain, pruritis, emotional concerns, embarrassment, anxiety, and interfere with activities of daily living, work activities, or interpersonal relations. To date, no data exist that compares quality of life outcomes - the fundamental metric to assess in an ambulatory dermatology population - between patients undergoing store and forward teledermatology consultations with patients managed by the conventional consult processes. Existing data does indicate that teledermatology is a reliable and accurate method of diagnosing skin disease.

Research Objectives - The purpose of this study was to compare store and forward teledermatology with a conventional clinic-based dermatology consultation process. Our primary objective was to determine whether the mean change in patient quality of life, as rated by the composite score and subscale scores of a skin-specific quality of life index (Skindex-16), differed between the time of randomization and 9 months for patients evaluated by store and forward teledermatology compared to conventional consult methods. Secondary objectives included (a) assessing quality of life between time of randomization and 3 months, (b) assessing time to initial definitive evaluation for patients using each modality, (c) evaluating clinical course using serial digital imaging, (d) comparing the costs and cost-effectiveness of store and forward teledermatology with conventional consult methods.

Project Methods - The study was a parallel-group, superiority, randomized clinical trial that compared store and forward teledermatology with a conventional clinic-based consult process. Patients were randomized using a simple randomization scheme stratified by site to one of the two consult modalities. Eligible patients included those being referred from the remote sites of primary care to the medical center-based sites of dermatology services. Skindex-16 was administered at baseline, 3 months, and 9 months. Time to initial definitive evaluation, calculated based on the need for and timing of a clinic-based visit was measured for both groups. Using digital images, clinical course was assessed on a 5 point scale by an expert panel of three dermatologists. Categories included resolved, improved, unchanged not clinically relevant, unchanged clinically relevant, and worse. Health care utilities were measured using time trade-off data and the Health Utilities Index Mark 2 (HUI2). We compared the costs of teledermatology with conventional consult methods by estimating the average cost per patient over the 9 month study period. Effectiveness was assessed using health care utilities and time to initial definitive evaluation. Costs were estimated from the VA perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single non-emergent skin condition being referred to a VA Dermatology Clinic
* Must be a veteran at the study site

Exclusion Criteria:

* Full body examination requested
* Unable to read or speak English
* Emergent skin condition
* Pending dermatology appointment within 9 months
* Previous enrollment in the study
* Impending move from the area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Whited, MD MHS, Principal Investigator — Harry S. Truman Memorial, Columbia, MO
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri

REFERENCES:
- [Background] Whited JD, Warshaw EM, Edison KE, Kapur K, Thottapurathu L, Raju S, Cook B, Engasser H, Pullen S, Parks P, Sindowski T, Motyka D, Brown R, Moritz TE, Datta SK, Chren MM, Marty L, Reda DJ. Effect of store and forward teledermatology on quality of life: a randomized controlled trial. JAMA Dermatol. 2013 May;149(5):584-91. doi: 10.1001/2013.jamadermatol.380. PMID 23426111
- [Result] Whited JD, Warshaw EM, Kapur K, Edison KE, Thottapurathu L, Raju S, Cook B, Engasser H, Pullen S, Moritz TE, Datta SK, Marty L, Foman NA, Suwattee P, Ward DS, Reda DJ. Clinical course outcomes for store and forward teledermatology versus conventional consultation: a randomized trial. J Telemed Telecare. 2013 Jun;19(4):197-204. doi: 10.1177/1357633x13487116. Epub 2013 May 23. PMID 23666440
- [Derived] Datta SK, Warshaw EM, Edison KE, Kapur K, Thottapurathu L, Moritz TE, Reda DJ, Whited JD. Cost and Utility Analysis of a Store-and-Forward Teledermatology Referral System: A Randomized Clinical Trial. JAMA Dermatol. 2015 Dec 1;151(12):1323-1329. doi: 10.1001/jamadermatol.2015.2362. PMID 26375589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 2008 and 2011.
Groups:
- Teledermatology Referrals: Store and forward teledermatology consult process
  Store and forward teledermatology: Standard electronic consult, standardized history, and image set
- Conventional Referrals: Conventional consult process
  Conventional consult process: Standard electronic consult
Period: Overall Study
Arm/Group | Teledermatology Referrals | Conventional Referrals
Started | 196 | 196
Completed | 160 | 166
Not Completed | 36 | 30
Not completed — Lost to Follow-up | 28 | 25
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Death | 2 | 1
Not completed — Misrandomization/Other Unspecified | 1 | 1

BASELINE CHARACTERISTICS:
Population: One patient assigned to teledermatology was misrandomized and not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teledermatology Referrals | Conventional Referrals | Total
Number analyzed (Participants) | 195 | 196 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.9) | 62.9 (13.9) | 62.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 190 | 192 | 382
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 193 | 191 | 384
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Skindex-16 Change Scores Between Baseline to Month 9 - Composite Score
Description: Skindex-16 Change Scores. Skindex-16 is a quality of life measure that assesses "bother." It includes the domains of symptoms, emotions, and functioning. A composite (total) score can also be calculated. The range of scores are 0 (never bothered) to 100 (always bothered) for subscale and composite scores. A negative change score represents a better quality of life. A change score of 10 points is considered clinically significant.
Time Frame: Baseline to Month 9
Population: Baseline to Month 9 Skindex-16 change scores - Composite Score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 164
units on a scale | -12.0 (24.5) | -13.2 (21.6)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

2. Secondary Outcome: Clinical Course Rating Between Baseline and Month 9
Description: Clinical course was assessed by review of serial digital images. The clinical course rating was provided by consensus opinion provided by a panel of three dermatologists that were not otherwise involved in the study. The rating categories were resolved, improved, unchanged - not clinically relevant, unchanged - clinically relevant, and worse.
Time Frame: Baseline to Month 9
Population: Clinical course rating between baseline and month 9
Measure: Number; unit: participants
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 125 | 136
participants
  Resolved | 31 | 35
  Improved | 59 | 63
  Unchanged - Not Clinically Relevant | 13 | 15
  Unchanged - Clinically Relevant | 13 | 17
  Worse | 9 | 6
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.88, Chi-squared

3. Primary Outcome: Skindex-16 Change Scores Baseline to Month 3 - Composite Score
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Baseline to Month 3 Skindex-16 change scores - Composite Score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 161 | 171
units on a scale | -7.8 (21.9) | -5.8 (19.1)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.39, t-test, 2 sided

4. Primary Outcome: Skindex-16 Change Scores Baseline to Month 9 - Symptoms Score
Description: as for outcome 1
Time Frame: Baseline to Month 9
Population: Baseline to Month 9 Skindex-16 change scores - Symptoms Score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 159 | 164
units on a scale | -10.3 (30.6) | -14.4 (28.2)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

5. Primary Outcome: Skindex-16 Changes Scores Baseline to Month 3 - Symptoms Score
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Baseline to Month 3 Skindex-16 change score - Symptoms Score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 171
units on a scale | -8.7 (29.8) | -8.0 (22.9)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.81, t-test, 2 sided

6. Primary Outcome: Skindex-16 Change Scores Between Baseline and Month 9 - Emotions Score
Description: as for outcome 1
Time Frame: Baseline to Month 9
Population: Baseline to Month 9 Skindex-16 change score - Emotions Score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 164
units on a scale | -19.7 (30.7) | -18.1 (25.1)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.61, t-test, 2 sided

7. Primary Outcome: Skindex-16 Change Scores Between Baseline to Month 3 - Emotions Score
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Baseline to Month 3 Skindex-16 change scores - Emotions Score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 171
units on a scale | -11.6 (27.2) | -8.9 (25.3)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

8. Primary Outcome: Skindex-16 Change Scores Between Baseline and Month 9 - Functioning Scores
Description: as for outcome 1
Time Frame: Baseline to Month 9
Population: Baseline to Month 9 Skindex-16 change scores - Functioning Scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 164
units on a scale | -6.0 (24.5) | -6.9 (22.3)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.73, t-test, 2 sided

9. Primary Outcome: Skindex-16 Change Scores Between Baseline and Month 3 - Functioning Score
Description: as for outcome 1
Time Frame: Baseline to Month 3
Population: Baseline to Month 3 Skindex-16 change scores - Functioning Scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 160 | 164
units on a scale | -3.2 (20.2) | -0.5 (20.9)
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

10. Secondary Outcome: Clinical Course Rating Between Baseline and First Clinic Visit
Description: as for outcome 2
Time Frame: Baseline to First Clinic Visit
Population: Clinical course rating between baseline and first clinic visit, if a visit occurred. Timeframe varied and only applied if a first clinic visit occurred.
Measure: Number; unit: participants
Arm/Group | Teledermatology Referrals | Conventional Referrals
Number analyzed (Participants) | 94 | 137
participants
  Resolved | 2 | 3
  Improved | 22 | 29
  Unchanged - Not Clinically Relevant | 10 | 20
  Unchanged - Clinically Relevant | 54 | 70
  Worse | 6 | 15
Statistical Analysis 1: Comparison: Teledermatology Referrals vs Conventional Referrals; Test type: Superiority or Other; p = 0.65, Chi-squared

ADVERSE EVENTS:
Arm/Group | Teledermatology Referrals | Conventional Referrals
Serious Adverse Events (participants affected / at risk) | 2/196 | 1/196
Other Adverse Events (participants affected / at risk) | 1/196 | 2/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teledermatology Referrals (N=196) | Conventional Referrals (N=196)
Death Unrelated to Study Participation (General disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teledermatology Referrals (N=196) | Conventional Referrals (N=196)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash from Sunscreen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection at Biopsy Site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes